CLINICAL TRIAL: NCT04448678
Title: Huntsman Intermountain Adolescent and Young Adult Cancer Care Program- Cancer Health Insurance Tool Study
Brief Title: Improving Health Insurance Experiences for Adolescent and Young Adult Cancer Patients
Acronym: HIAYA CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other); Massachusetts General Hospital (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anne Kirchhoff, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB_00127029; 1R01CA242729-01 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Adolescent; Young Adult; Cancer
Keywords: Education; Insurance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know who is receiving additional health insurance navigation or standard navigation. The outcome assessor will also be blinded to which participants received health insurance navigation. Blinding for the outcome assessor will be kept throughout the entirety of the analysis. Groups will be identified for analysis with ambiguous categories such as group 1 and group 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIEP intervention (Experimental): Participants will be randomized to receive the insurance navigation intervention from patient navigators, which includes four, one hour long, educational learning sessions. Randomization will be done by age at diagnosis and site.
  Interventions: Behavioral: Health Insurance Education Program (HIEP)
- Usual Care (Active Comparator): Participants will be randomized to receive standard navigation provided by patient navigators ("usual care").
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Health Insurance Education Program (HIEP) — [See arm/group descriptions]
  Arms: HIEP intervention
Other: Usual Care — [See arm/group descriptions]
  Arms: Usual Care

SUMMARY:
This is a test of an existing health insurance education program (HIEP) in adolescent and young adult (AYA) individuals (aged 18-39) diagnosed with cancer. The study will evaluate whether the HIEP delivered by patient navigators improves participants' health insurance and cost-related literacy compared to usual navigation care, which does not include education on insurance and medical costs. The study team hypothesizes that: The HIEP will improve participants' health insurance and cost-related literacy compared to usual navigation care. Specifically, that participants in the intervention arm will report greater 1) health insurance and cost literacy, including confidence with provider communication about costs, 2) familiarity with ACA policies, and 3) improvement in financial distress related to medical costs. Participants will fill out a survey upon enrollment and a follow up survey 3 months after meeting with a patient navigator where they may or may not receive the HIEP.

DETAILED DESCRIPTION:
The goal of this research is to refine and pilot test an existing health insurance education program (HIEP) to improve health insurance and cost-related literacy among adolescent and young adult (AYA) individuals who have recently been diagnosed with cancer. This study will be conducted within the Huntsman-Intermountain Adolescent and Young Adult (HI-AYA) Cancer Care Program, which is a unique collaboration between the Huntsman Cancer Institute and Intermountain Healthcare, the largest oncology providers in Utah. Initially, age-related differences related to health insurance and cost literacy among AYAs diagnosed with cancer ages 18-26 and 27-39 years will be identified, and the HIEP materials will be adapted accordingly. The HIEP delivered by the HI-AYA patient navigators, will be investigated to see if it improves participants' health insurance and cost-related literacy.

Upon enrollment, participants will fill out a survey containing questions about their current health insurance plan, financial status, demographics, health insurance knowledge, and financial toxicity. Participants will then be randomized into separate trial arms after which participants in both groups will meet with a HI-AYA patient navigator. Participants in the interventional arm will receive 4 educational sessions surrounding health insurance use and laws (four sessions total occurring approximately every two weeks). These educational sessions will be conducted, in person, over video conference calls, or over the telephone, and will cover:

* health insurance terms and concepts
* insurance coverage (insurance cards, bills, schedule and explanation on benefits)
* health insurance laws, rights and the appeals process
* budgeting and resources. These sessions will be scheduled with each participant according to their availability, with the goal of meeting every other week.

Approximately three months after meeting with the patient navigator, participants in both arms of the trial will fill out a second survey, including similar questions to those in the first survey as well as questions surrounding satisfaction with the HIEP and the patient navigator delivery for those who received the HIEP. After the post survey is complete, a small subset of participants in both the intervention and control arm will be randomly selected to complete an interview to better understand satisfaction with patient navigation, the intervention, recommendations for modifications on delivery modality, and recommendations for intervention topics and content modifications to identify components of the HIEP that require refinement prior to potential scaling of the intervention to a larger sample. Another small subset of participants will be randomly selected to complete an interview from the control arm to discuss their satisfaction with their patient navigation and to ask how they found resources concerning health insurance during their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Were diagnosed with cancer between the ages of 18 and 39 AND
* Are within 1 year of a cancer diagnosis AND
* Are actively receiving chemotherapy, surgery, radiation, and/or hormonal therapy AND
* Are currently insured AND
* A patient at Primary Children's Hospital, Intermountain Medical Center or Huntsman Cancer Institute AND
* Speak English AND
* Have access to an electronic device compatible with video conferencing (e.g., smartphone, laptop, etc.).

Exclusion Criteria:

* Are unable to participate due to developmental delay OR
* Speak a language other than English OR
* Are currently uninsured OR
* Do not have access to an electronic device compatible with video conferencing (e.g., smartphone, laptop, etc.).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Kirchhoff, PhD, MPH, Principal Investigator — University of Utah Department of Pediatrics
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaca Lopez PL, Warner EL, Waters AR, van Thiel Berghuijs KM, Anderson JS, Ray N, Tsukamoto T, Kaddas HK, Fair D, Lewis M, Park ER, Perez GK, Kirchhoff AC. Adaptation and Development of a Health Insurance Education Program for Adolescent and Young Adult Cancer Patients. J Adolesc Young Adult Oncol. 2023 Oct;12(5):692-700. doi: 10.1089/jayao.2022.0103. Epub 2023 Jan 27. PMID 36706435
- [Derived] Mann K, Waters AR, Park ER, Perez GK, Vaca Lopez PL, Kaddas HK, Warner EL, Ray N, Tsukamoto T, Allen K, Haaland B, Fair DB, Lewis MA, Kirchhoff AC. HIAYA CHAT study protocol: a randomized controlled trial of a health insurance education intervention for newly diagnosed adolescent and young adult cancer patients. Trials. 2022 Aug 19;23(1):682. doi: 10.1186/s13063-022-06590-5. PMID 35986416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We decided to overshoot our original target just to have the extra data.
Period: Overall Study
Arm/Group | HIEP Intervention | Usual Care
Started | 45 | 41
Completed | 25 | 39
Not Completed | 20 | 2

BASELINE CHARACTERISTICS:
Population: Insured cancer patients between the ages of 18-39 who are within their first year of treatment at Huntsman Cancer Institute or the Intermountain Network.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIEP Intervention | Usual Care | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 41 | 86
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.96 (7.19) | 28.71 (6.15) | 28.84 (6.68)
Age, Customized [Count of Participants; unit: Participants]
  Younger Group Age 18-25 | 17 | 13 | 30
  Older Group Age 26-39 | 28 | 28 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 39 | 30 | 69
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 26 | 62
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  United States | 45 | 41 | 86
COmprehensive Score for financial Toxicity (COST) [Mean (Standard Deviation); unit: Score on a scale] — The COST Score is a validated patient reported outcome measure which screens for financial toxicity in cancer patients. Lower scores indicate increased financial toxicity or worse outcomes. Scores range from 0-44. Population: Some of the participants (n=4) did not fill in all of the fields required for us to analyze their COST score.
  Score on a scale
    number analyzed (Participants) | 43 | 39 | 82
    (all) | 19.72 (9.72) | 20.18 (12.20) | 19.94 (10.90)
Health Insurance Literacy Measure (HILM) [Mean (Standard Deviation); unit: Score on a scale] — The HILM is a validated measure that assess a patients health insurance literacy and which areas a patient may need additional assistance with insurance issues. Traditionally, the measure consists of 4 categories, confidence choosing health insurance, comparing health plans, confidence using health insurance and being proactive with health insurance. For this study, we focused on sections concerning confidence using health insurance and being proactive with health insurance. Scores range from 9-36. Lower scores indicate lower health insurance literacy and worse outcomes. Population: Some of the participants (n=1) did not fill in all of the fields required for us to analyze their HILM score.
  Score on a scale
    number analyzed (Participants) | 44 | 41 | 85
    (all) | 22.64 (5.21) | 22.46 (5.81) | 22.55 (5.48)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Measurement
Description: Comparing total number of individuals enrolled and randomized vs completed study (completion of both surveys for control or both surveys and all of the sessions for intervention.)
Time Frame: Post-Assessment survey (Weeks 13 (+/- 2 weeks))
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Number of participants who were randomized into care as usual versus those who completed the study (follow up survey).
- HIEP Intervention: Number of participants who were randomized into the Health Insurance Educational Program versus those who completed the study (all 4 sessions and the follow up survey).
Arm/Group | Usual Care | HIEP Intervention
Number analyzed (Participants) | 41 | 45
Participants | 39 | 25

2. Primary Outcome: Acceptability - Module Satisfaction
Description: Questions surrounding satisfaction with the HIEP. These will be asked at the post-assessment interview and will consist of participants responses surrounding satisfaction with the HIEP. We will report percentages of participants who did 1 or more session and reported satisfaction with the HIEP.
Time Frame: Post-Assessment interview (Weeks 18 (+/- 2 weeks))
Population: Analysis of participants satisfaction from questions asked in the exit interview. Only including participants who were randomized into the intervention, then the exit interviews, and completed at least one session of the HIEP.
Measure: Count of Participants; unit: Participants
Groups:
- HIEP Intervention: Participants will be randomized to receive the insurance navigation intervention from patient navigators, which includes four, 30-45 minute long, educational learning sessions. Randomization will be done by age at diagnosis and site. Those intervention participants will be randomized into exit interviews where we will get the data about satisfaction with the HIEP.
Arm/Group | HIEP Intervention | Usual Care
Number analyzed (Participants) | 10 | 0
Participants | 10 | 0

3. Primary Outcome: Navigator Satisfaction
Description: Validated Patient Satisfaction with Navigator Interpersonal Relationship (PSN-I) measure at post assessment survey. This score ranges from 0-45 with higher scores indicating higher satisfaction. We will report the mean and standard deviation.
Time Frame: Post-Assessment survey (Weeks 13 (+/- 2 weeks))
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIEP Intervention | Usual Care
Number analyzed (Participants) | 45 | 41
score on a scale | 30.84 (16.15) | 30.32 (12.95)

4. Secondary Outcome: Changes in Efficacy- Health Insurance Literacy
Description: Differences between Health Insurance Literacy Measure (HILM) reported at the intro baseline and exit post-assessment survey. For this study, the last two sections (3&4) of the HILM were used. Scores range from 9-36 with lower scores indicate lower health insurance literacy and worse outcomes. Differences will be examined by age group and by treatment arm. We report mean and standard deviation. Please note that not all participants, filled out all necessary questions at both timepoints to be assessed.
Time Frame: Baseline (Week 0) and Post Assessment survey (Weeks 13 (+/- 2 weeks))
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Combined: All participants
Arm/Group | HIEP Intervention | Usual Care | Combined
Number analyzed (Participants) | 36 | 36 | 72
Score on a scale | 5.39 (6.44) | 2.30 (6.06) | 3.84 (6.40)
Statistical Analysis 1: Comparison: HIEP Intervention vs Usual Care; Test type: Other; p = 0.0401, t-test, 2 sided

5. Secondary Outcome: Changes in Efficacy- Affordable Care Act (ACA) Familiarity
Description: Questions surrounding familiarity with the ACA reported at the baseline and post-assessment survey. Values range from 0 to 28 with higher scores indicating better familiarity with ACA concepts. We will report the mean and standard deviation of the difference in response scores between baseline and post assessment for the control and intervention. Please note that not all participants, filled out all necessary questions at both timepoints to be assessed.
Time Frame: Baseline (Week 0) and Post Assessment survey (Weeks 13 (+/- 2 weeks))
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HIEP Intervention | Usual Care | Combined
Number analyzed (Participants) | 37 | 37 | 74
Score on a scale | 5.84 (6.30) | 2.03 (4.89) | 3.93 (5.92)
Statistical Analysis 1: Comparison: HIEP Intervention vs Usual Care; Test type: Other; p = 0.0049, t-test, 2 sided

6. Secondary Outcome: Changes in Efficacy-Financial Distress
Description: Differences between COmprehensive Score for financial Toxicity (COST) reported at the baseline and post-assessment survey. Values range from 0 to 44 where lower COST scores indicate worse financial toxicity. Differences will be examined by age group and by treatment arm. We will report mean and standard deviation. Please note that not all participants, filled out all necessary questions at both timepoints to be assessed.
Time Frame: Baseline (Week 0) and Post Assessment survey ( Weeks 13 (+/- 2 weeks))
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HIEP Intervention | Usual Care | Combined
Number analyzed (Participants) | 35 | 36 | 71
Score on a scale
  Younger group (18-25) | 3.70 (9.59) | 2.89 (9.44) | 3.32 (9.26)
  Older group (26-39) | 3.08 (8.45) | 0.741 (6.42) | 1.87 (7.48)
  Combined (18-39) | 3.25 (8.65) | 1.28 (7.20) | 2.25 (7.95)
Statistical Analysis 1: Comparison: HIEP Intervention vs Usual Care; Test type: Other; p = 0.297, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored for this study;.
Description: As this study was an educational intervention on health insurance, mortality, serious and non-serious adverse events were not monitored/assessed.
Arm/Group | HIEP Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT04448678/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT04448678/SAP_003.pdf
  • Informed Consent Form: UniversityofUtah (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT04448678/ICF_000.pdf
  • Informed Consent Form: IntermountainHealthCare (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04448678/ICF_001.pdf